CLINICAL TRIAL: NCT06968364
Title: Evaluation of the Safety and the Preterm Birth Predictive Capacity of the Clinical Investigation Device 'Cervisense TPTL': an International Clinical Study
Brief Title: FB-CT2 Includes Two Prospective, Multi-centre Studies With a Medical Device in Hospital Settings: a Randomized, Dual-arm, Open-label Pilot Study in Spain, Followed by a Single-arm, Non-randomized, Open-label International Pivotal Study
Acronym: FB-CT2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ultrasound-Innovation Medtech, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: FB-CT2
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Threatened Preterm Labor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervisense (Experimental): Cervisense arm: Cervisense Intravaginal Probe V0.1 cervical stiffness evaluation.
  Interventions: Device: Cervisense Intravaginal Probe V0.1 cervical stiffness evaluation.
- Control arm (only in Pilot Phase) (Active Comparator): Control arm: Cervicometry measured with transvaginal ultrasound
  Interventions: Device: Transvaginal ultrasound

INTERVENTIONS:
Device: Cervisense Intravaginal Probe V0.1 cervical stiffness evaluation. — The Cervisense Intravaginal Probe V0.1 measures cervical stiffness. It is an in-vivo predictive technology that, by using torsional waves, quantifies the mechanical properties (specifically the shear modulus, or resistance of the cervix to shear deformation (kPa), of cervical tissue with extremely high precision. Torsional wave is a type of mechanical wave characterized by a rotational motion and low energy levels (it uses 1000 times less energy than other mechanical waves such as ultrasound). These waves propagate through the tissue, and their propagation speed, which is related to the stiffness (waves propagate faster in stiffer tissues), is measured using piezoelectric sensors.
  Arms: Cervisense
Device: Transvaginal ultrasound — Cervicometry measured with transvaginal ultrasound
  Arms: Control arm (only in Pilot Phase)

SUMMARY:
The goal of this clinical trial is to evaluate the safety and the ability of a clinical investigation device (Cervisense TPTL) to predict the risk of spontaneous preterm birth in pregnant women with symptoms of threatened preterm labor (TPTL), between 28+0 and 36+6 weeks of gestation. The main questions it aims to answer are:

Does the Cervisense TPTL device predict spontaneous preterm birth within 7 days?

Is the device safe and technically reliable in a hospital setting?

Researchers will conduct a Pilot Study (randomized, dual-arm) followed by a Pivotal Study (single-arm) to assess technical feasibility and predictive performance.

Participants will undergo an intravaginal measurement of cervical stiffness using the Cervisense Intravaginal Probe. They will be followed for 14 days after the assessment to record delivery outcomes and any adverse events.

DETAILED DESCRIPTION:
The study titled "Evaluation of the safety and the preterm birth predictive capacity of the clinical investigation device 'Cervisense TPTL': an international clinical study" is designed to assess both the safety and performance of the Cervisense TPTL device in predicting spontaneous preterm birth. It is being conducted across various Gynaecology, Obstetrics, and Emergency Services in hospitals throughout Spain and Germany.

Cervisense TPTL is the investigational product being evaluated. It includes two components: the Cervisense Intravaginal Probe V0.1, which measures cervical stiffness, and the Fine Birth algorithm, which combines the measurement with clinical data to assess the short-term risk of spontaneous preterm labor.

The device is intended for use in pregnant women showing symptoms of threatened preterm labor (TPTL), with intact amniotic membranes and a single fetus, between 28 weeks and 36 weeks plus 6 days of gestation. Its purpose is to determine the risk of spontaneous preterm birth within the following 7 days.

The clinical investigation is structured in two phases. The pilot study is a randomized, dual-arm, open-label, interventional, multi-centre study conducted in Spain. Participants are randomized 1:1 to receive either the standard of care or the Cervisense evaluation. The pivotal study is non-randomized and single-arm, also open-label and interventional, conducted at a larger scale across multiple centres in both Spain and Germany.

The main goal is to confirm that the device is safe to use and reliable in clinical settings. For safety, all adverse events associated with the use of the device are documented and analyzed in terms of severity, duration, and required intervention. Special attention is given to potential complications such as tissue trauma or infection. To ensure unbiased evaluation, a Clinical Events Committee and a Data Safety Monitoring Board have been established to independently review adverse events and guide study continuation.

Inclusion Criteria:

* Female ≥18 years
* Singleton pregnancy
* Live fetus, 28w+0d-36w+6d GA
* Intact membranes
* Cervical dilatation <2 cm
* Signed informed consent
* Regular uterine contractions (≥8/60 min) (Pivotal only)

Exclusion Criteria:

* Latex allergy
* Prolapsed membranes
* Fetal malformation
* Fetal infection
* Vaginal bleeding (severe or persistent)
* Cervical cerclage
* Müllerian anomalies
* Pessary use
* Regular uterine contractions (reported by patient) (Pilot only)
* History of preterm birth or TPTL (Pilot only)
* Vasa/placenta previa (Pilot only)
* Gastrointestinal or urinary infections (Pivotal only)

ELIGIBILITY:
Inclusion Criteria:

* Female ≥18 years
* Singleton pregnancy
* Live fetus, 28w+0d-36w+6d GA
* Intact membranes
* Cervical dilatation <2 cm
* Signed informed consent
* Regular uterine contractions (≥8/60 min) (Pivotal only)

Exclusion Criteria:

* Latex allergy
* Prolapsed membranes
* Fetal malformation
* Fetal infection
* Vaginal bleeding (severe or persistent)
* Cervical cerclage
* Müllerian anomalies
* Pessary use
* Regular uterine contractions (reported by patient) (Pilot only)
* History of preterm birth or TPTL (Pilot only)
* Vasa/placenta previa (Pilot only)
* Gastrointestinal or urinary infections (Pivotal only)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women with singleton gestation between 28w+0d and 36w+6d.
Enrollment: 457 (Estimated)
Dates: Start 2025-05-10 (Estimated); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
≥90% Specificity and ≥50% Sensitivity for predicting spontaneous preterm birth within 7 days (Pivotal Phase) | From enrollment until delivery
  It will be determined in terms of accuracy, specifically with Specificity and Sensitivity as primary endpoints. Cervisense TPTL will be considered effective in screening for preterm birth risk if the validation study demonstrates at least 90% Specificity and 50% Sensitivity in detecting spontaneous preterm birth within the next 7 days of the cervical stiffness measurement among pregnant women with gestational age between 28w+0d and 36w+6d with suspected and symptomatic Threatened Preterm Labor (TPTL) presenting to the emergency department.
Document and analyse all adverse events related to device use (severity, duration, intervention) (Pilot and Pivotal Phases) | From enrollment until delivery
  To document and analyse all adverse events related to the device use, categorized by severity, duration, and required intervention. Exhaustive monitoring of complications directly attributable to the device or its usage, such as tissue damage or active infection.
Technical problems ratio (Pilot Phase) | From enrollment until the use of the device
  To report less than 10 technical problems that impeded the physician from performing cervical stiffness measurements
Probe repeatability (Pilot Phase) | From enrollment until the use of the device
  To have an average repeatability rate greater than 75%
Valid measurements obtained (Pilot Phase) | From enrollment until the use of the device
  To achieve more than 80% of valid cases among the measures obtained

SECONDARY OUTCOMES:
Monitor labour progression indicators (Pilot and Pivotal Phases) | From enrollment until the 14-days follow-up
  To monitor key indicators of labour progression, such as frequency and intensity of contractions, and foetal descent after using the device to determine based on clinical criteria if there are any significant changes in labour progression indicators that could be attributed to its use.
Monitor trauma indicators (e.g., petechiae, bleeding) (Pilot and Pivotal Phases) | From enrollment until the 14-days follow-up
  To monitor key indicators of potential trauma caused by the device entering the vagina or contacting the cervix, such as bruising (petechiae) or bleeding. Visual evaluation of the vagina and the cervix will be performed before and immediately after the use of the device and any significant changes that could be attributed to its use will be documented.
VAS pain score ≤3 (mild/no pain) (Pilot and Pivotal Phases) | From enrollment until the use of the device
  To achieve a VAS score attributed to the use of Cervisense Intravaginal Probe V0.1 m≤ 3, which is equivalent to mild or no pain.
Specificity, Sensitivity, PPV, NPV within 10 and 14 days (Pivotal Phase) | From enrollment until delivery
  To estimate and report Cervisense TPTL Specificity, Sensitivity, Positive predictive value (PPV) and Negative predictive value (NPV) in screening for spontaneous preterm birth within the next 10 and 14 days of the cervical stiffness measurement among pregnant women with gestational age between 28w+0d and 36w+6d with suspected and symptomatic Threatened Preterm Labour (TPTL) presenting to the emergency department.
Subgroup analysis (gestational age, obstetric history) (Pivotal Phase) | From enrollment until delivery
  To estimate and report Cervisense TPTL Specificity, Sensitivity, Positive predictive value (PPV) and Negative predictive value (NPV) in screening for spontaneous preterm birth within the next 14 days of the cervical stiffness measurement among pregnant women with gestational age between 28w+0d and 36w+6d with suspected and symptomatic Threatened Preterm Labour (TPTL) presenting to the emergency department.
Training performance (Pivotal Phase) | From enrollment until delivery
  To evaluate the performance of the device in different subgroups (gestational age, previous pregnancies, previous deliveries previous miscarriages, previous episode of TPTL).
Operator satisfaction (SUS) (Pilot and Pivotal Phases) | From enrollment until the use of the device
  To measure the operator degree of satisfaction with the Cervisense technique with the SUS (System Usability Scale).
Comparison with PartoSure and cervical length (at 7, 10, 14 days) (Pivotal Phase) | From enrollment until delivery
  To compare the Specificity, Sensitivity, Positive predictive value (PPV) and Negative predictive value (NPV) of Cervisense TPTL with the ones obtained with PartoSure test and cervical length within the next 7, 10 and 14 days of the cervical stiffness measurement among pregnant women with gestational age between 28w+0d and 36w+6d with suspected and symptomatic Threatened Preterm Labour (TPTL) presenting to the emergency department.
Degree of success obtained during the use of the Cervisense Intravaginal Probe (Pilot Phase) | From enrollment until the use of the device
  To measure the degree of success obtained during the use of Cervisense Intravaginal Probe V0.1: device ID, operator profile and code, number of repetitions, % repeatability of the measurement, incidents and probe cover breakage

CONTACTS AND LOCATIONS:
Locations (14):
- Spain (14):
  - H. Universitario de A Coruña, A Coruña
  - H. Clínic de Barcelona, Barcelona
  - H. Sant Joan de Déu, Barcelona
  - H. Vall d'Hebron, Barcelona
  - H. Universitario de Basurto, Bilbao
  - H. Universitario de Cruces, Bilbao
  - H. Universitario de Donostia, Donostia / San Sebastian
  - H. Universitario San Cecilio, Granada
  - H. Materno Infantil de Gran Canaria, Las Palmas de Gran Canaria
  - H. General Universitario Gregorio Marañón, Madrid
  - H. Universitario de Torrejón, Madrid
  - H. Universitario La Paz, Madrid
  - H. Universitario de Málaga, Málaga
  - H. Virgen Arrixaca, Murcia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Papiernik E, Bouyer J, Collin D, Winisdoerffer G, Dreyfus J. Precocious cervical ripening and preterm labor. Obstet Gynecol. 1986 Feb;67(2):238-42. doi: 10.1097/00006250-198602000-00014. PMID 3945433
- [Background] Parra-Saavedra M, Gomez L, Barrero A, Parra G, Vergara F, Navarro E. Prediction of preterm birth using the cervical consistency index. Ultrasound Obstet Gynecol. 2011 Jul;38(1):44-51. doi: 10.1002/uog.9010. PMID 21465603
- [Background] Molina FS, Pardo L, Munoz MD, Aiartzaguena A, Valladolid A, Blanco JE, Burgos J, Gil MM. Reproducibility and usability assessment of the novel Fine Birth device for threatened preterm labor diagnosis. Am J Obstet Gynecol MFM. 2023 Jul;5(7):100982. doi: 10.1016/j.ajogmf.2023.100982. Epub 2023 Apr 23. PMID 37094638
- [Background] Melchor JC, Navas H, Marcos M, Iza A, De Diego M, Rando D, Melchor I, Burgos J. Predictive performance of PAMG-1 vs fFN test for risk of spontaneous preterm birth in symptomatic women attending an emergency obstetric unit: retrospective cohort study. Ultrasound Obstet Gynecol. 2018 May;51(5):644-649. doi: 10.1002/uog.18892. Epub 2018 Mar 26. PMID 28850753
- [Background] Melchor JC, Khalil A, Wing D, Schleussner E, Surbek D. Prediction of preterm delivery in symptomatic women using PAMG-1, fetal fibronectin and phIGFBP-1 tests: systematic review and meta-analysis. Ultrasound Obstet Gynecol. 2018 Oct;52(4):442-451. doi: 10.1002/uog.19119. Epub 2018 Sep 4. PMID 29920825
- [Background] Masso P, Callejas A, Melchor J, Molina FS, Rus G. In Vivo Measurement of Cervical Elasticity on Pregnant Women by Torsional Wave Technique: A Preliminary Study. Sensors (Basel). 2019 Jul 24;19(15):3249. doi: 10.3390/s19153249. PMID 31344796
- [Background] Jackson GM, Ludmir J, Bader TJ. The accuracy of digital examination and ultrasound in the evaluation of cervical length. Obstet Gynecol. 1992 Feb;79(2):214-8. doi: 10.3109/01443619209013646. PMID 1731287
- [Background] Horinouchi T, Yoshizato T, Muto M, Fujii M, Kozuma Y, Shinagawa T, Morokuma S, Kakuma T, Ushijima K. Gestational age-related changes in shear wave speed of the uterine cervix in normal pregnancy at 12-35 weeks' gestation. J Perinat Med. 2019 May 27;47(4):393-401. doi: 10.1515/jpm-2018-0250. PMID 30817303
- [Background] Holcomb WL Jr, Smeltzer JS. Cervical effacement: variation in belief among clinicians. Obstet Gynecol. 1991 Jul;78(1):43-5. PMID 2047066
- [Background] Goldenberg RL, Mercer BM, Meis PJ, Copper RL, Das A, McNellis D. The preterm prediction study: fetal fibronectin testing and spontaneous preterm birth. NICHD Maternal Fetal Medicine Units Network. Obstet Gynecol. 1996 May;87(5 Pt 1):643-8. doi: 10.1016/0029-7844(96)00035-x. PMID 8677060
- [Background] Carlson LC, Feltovich H, Palmeri ML, Dahl JJ, Munoz del Rio A, Hall TJ. Estimation of shear wave speed in the human uterine cervix. Ultrasound Obstet Gynecol. 2014 Apr;43(4):452-8. doi: 10.1002/uog.12555. Epub 2014 Mar 12. PMID 23836486
- [Background] Callejas A, Gomez A, Faris IH, Melchor J, Rus G. Kelvin-Voigt Parameters Reconstruction of Cervical Tissue-Mimicking Phantoms Using Torsional Wave Elastography. Sensors (Basel). 2019 Jul 25;19(15):3281. doi: 10.3390/s19153281. PMID 31349721
- [Background] BISHOP EH. PELVIC SCORING FOR ELECTIVE INDUCTION. Obstet Gynecol. 1964 Aug;24:266-8. No abstract available. PMID 14199536